CLINICAL TRIAL: NCT01357720
Title: A Phase IV, Single-blind, Randomized, Controlled, Monocentric Study to Assess the Interchangeability of Quinvaxem (DTwP-HepB-Hib) as the 2nd and 3rd Dose After Initial Vaccination With Tritanrix HB+Hib (DTwP-HepB/Hib) With Respect to Safety and Immunogenicity in Healthy Infants at 6, 10 and 14 Weeks of Age
Brief Title: Study to Assess if Quinvaxem Can be Interchanged With Other Pentavalent Vaccines During Standard Childhood Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QVX-V-A001
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Diphtheria; Pertussis; Tetanus; Hepatitis B; Haemophilus Infections
Keywords: Vaccination; Immunisation; Virus; Diphtheria; Pertussis; Tetanus; Hepatitis B; Haemophilus Influenzae; Immunity
MeSH Terms: conditions — Diphtheria; Whooping Cough; Tetanus; Hepatitis B; Haemophilus Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quinvaxem (Experimental)
  Interventions: Biological: Quinvaxem
- Tritanrix Hib/HepB + Quinvaxem (Active Comparator)
  Interventions: Biological: Quinvaxem/Tritanrix

INTERVENTIONS:
Biological: Quinvaxem — A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), whole-cell inactive pertussis bacteria (>= 4 IU), 10 mcg Hib oligosaccharide conjugate (approx. 25 mcg CRM197), 10 mcg Hepatitis B surface antigen
  One dose of Quinvaxem given at Weeks 6, 10 and 14
  Arms: Quinvaxem
Biological: Quinvaxem/Tritanrix — A single dose (0.5 mL) of Quinvaxem contains:
  diphtheria antitoxin (>= 30 IU), tetanus antitoxin (>= 60 IU), inactive pertussis bacteria (>= 4 IU), 10 mcg Hib polysaccharide conjugate (approx. 25 mcg tetanus toxoid), 10 mcg Hepatitis B surface antigen
  One dose of Quinvaxem given at Weeks 6, 10 and 14
  Arms: Tritanrix Hib/HepB + Quinvaxem

SUMMARY:
This is a study to show that vaccination with 1 dose of Tritanrix HB+Hib followed by Quinvaxem vaccine as the 2nd and 3rd dose is not inferior to vaccination with Quinvaxem for all 3 doses, with respect to protection against all antibodies (anti-hepatitis B surface antibodies, anti-polyribosyl ribitol phosphate (PRP), anti-diphtheria, anti-tetanus and anti-Bordetella pertussis) 1 month after completion of the 6-10-14 week vaccination course.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 42 and 64 days of age at the time of the first vaccination
* Written informed consent obtained from parents/legal guardian of the subject
* Free of obvious health problems as established by medical history and/or clinical examination before entering the study
* Hepatitis B vaccination at birth (within 48 hours) Available for all scheduled study visits

Exclusion Criteria:

* Use of any investigational drug or any investigational vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and safety follow-up
* Planned administration of a vaccine not foreseen by the study protocol
* Known or suspected impairment of immune function, known Human immunodeficiency virus (HIV)-positivity, receiving immunosuppressive therapy, or having received systemic immunosuppressive therapy within 1 month prior to study entry (note: inhaled and topical steroids are allowed)
* Administration of parenteral immunoglobulin preparation and/or blood products since birth
* Previous vaccination against Haemophilus influenzae type b (Hib) and/or diphtheria, tetanus, pertussis (DTP)
* History of anaphylaxis, or any serious vaccine reaction, or allergy to any vaccine component or to products containing mercury compounds, such as sodium ethylmercuro-thiosalicylate
* Significant acute infection
* Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
* Participation in another clinical study

Ages: 42 Days to 64 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria RZ Capeding, MD, Principal Investigator — Research Institute for Tropical Medicine (RITM)
Locations (1):
- Research Institute for Tropical Medicine, City of Muntinlupa, Philippines

REFERENCES:
- [Derived] Capeding MR, Jica C, Macura-Biegun A, Rauscher M, Alberto E. Interchangeability of Quinvaxem during primary vaccination schedules: results from a phase IV, single-blind, randomized, controlled, single-center, non-inferiority study. Vaccine. 2014 Feb 7;32(7):888-94. doi: 10.1016/j.vaccine.2013.10.059. Epub 2013 Oct 29. PMID 24176498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at two vaccination sites in the Philippines:
  First subject first visit (FSFV): 30 May 2011 Last subject last visit (LSLV): 30 September 2011
Groups:
- Quinvaxem: Three-dose schedule: 6, 10 and 14 weeks of age Weeks 6, 10 and 14: single doses of Quinvaxem
- Tritanrix Hib/HepB + Quinvaxem: Three-dose schedule: 6, 10 and 14 weeks of age Week 6: single dose of Tritanrix HB+Hib Weeks 10 and 14: single doses of Quinvaxem
Period: Overall Study
Arm/Group | Quinvaxem | Tritanrix Hib/HepB + Quinvaxem
Started | 200 | 200
Completed | 198 | 195
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quinvaxem | Tritanrix Hib/HepB + Quinvaxem | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 200 | 200 | 400
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: weeks] | 6.8 (0.91) | 6.7 (0.86) | 6.7 (0.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 105 | 206
  Male | 99 | 95 | 194

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Rate: Anti-PRP Antibodies
Description: Percentage of subjects with an anti-PRP titer ≥0.15 µg/mL (i.e. seroprotection rate)
Time Frame: 1 month after the third vaccination
Population: Available observations at Visit 4
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Quinvaxem | Tritanrix Hib/HepB + Quinvaxem
Number analyzed (Participants) | 197 | 193
percentage of subjects | 100 [98.1 to 100] | 100 [98.1 to 100]

2. Primary Outcome: Seroprotection Rate: Anti-hepatitis B Surface Antibodies
Description: Percentage of subjects with an anti-hepatitis B surface antibody titer ≥10 IU/L (i.e. seroprotection rate)
Time Frame: 1 month after the third vaccination
Population: Available observations at Visit 4
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Quinvaxem | Tritanrix Hib/HepB + Quinvaxem
Number analyzed (Participants) | 198 | 194
percentage of subjects | 94.9 [90.9 to 97.6] | 97.4 [94.1 to 99.2]

3. Primary Outcome: Seroprotection Rate: Anti-diphtheria Toxoid Antibodies
Description: Percentage of subjects with antibody levels against diphtheria toxoid ≥0.1 IU/mL (i.e. seroprotection rate)
Time Frame: 1 month after the third vaccination
Population: Available observations at Visit 4
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Quinvaxem | Tritanrix Hib/HepB + Quinvaxem
Number analyzed (Participants) | 198 | 194
percentage of subjects | 99.5 [97.2 to 100] | 100 [98.1 to 100]

4. Primary Outcome: Seroprotection Rate: Anti-tetanus Toxoid Antibodies
Description: Percentage of subjects with antibody levels against tetanus toxoid ≥0.1 IU/mL (i.e. seroprotection rate)
Time Frame: 1 month after the third vaccination
Population: Available observations at Visit 4
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Quinvaxem | Tritanrix Hib/HepB + Quinvaxem
Number analyzed (Participants) | 198 | 194
percentage of subjects | 100 [98.2 to 100] | 100 [98.1 to 100]

5. Primary Outcome: Seroprotection Rate: Anti-B. Pertussis Antibodies
Description: Percentage of subjects with an anti-B. pertussis antibody titer ≥20 EU/mL or a 4-fold increase over baseline (i.e. seroconversion rate)
Time Frame: 1 month after the third vaccination
Population: Available observations at Visit 4
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Quinvaxem | Tritanrix Hib/HepB + Quinvaxem
Number analyzed (Participants) | 198 | 194
percentage of subjects | 99.0 [96.4 to 99.9] | 100 [98.1 to 100]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic AEs were collected on the day of vaccination, and for the four days after the day of each vaccination. Unsolicited AEs were collected at each study visit up to Day 85.
Arm/Group | Quinvaxem | Tritanrix Hib/HepB + Quinvaxem
Serious Adverse Events (participants affected / at risk) | 0/200 | 2/200
Other Adverse Events (participants affected / at risk) | 180/200 | 180/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinvaxem (N=200) | Tritanrix Hib/HepB + Quinvaxem (N=200)
Viral encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinvaxem (N=200) | Tritanrix Hib/HepB + Quinvaxem (N=200)
Injection site pain (General disorders) | 137 (293) | 157 (338)
Injection site induration (General disorders) | 74 (138) | 82 (145)
Injection site erythema (General disorders) | 59 (87) | 54 (73)
Pyrexia (General disorders) | 88 (133) | 95 (137)
Upper respiratory tract infection (Infections and infestations) | 46 (55) | 54 (69)
Nasopharyngitis (Infections and infestations) | 7 (7) | 9 (10)
Rhinitis (Infections and infestations) | 7 (8) | 7 (7)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any material for public dissemination will be submitted to the Sponsor for review at least ninety (90) days prior to submission for publication, public dissemination, or review by a publication committee